CLINICAL TRIAL: NCT00809939
Title: 17 Alfa Hydroxyprogesterone Caproate Versus Natural Progesterone for the Prevention of Preterm Labor
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0129-08-MMC Ver:1
Record Dates: First submitted 2008-12-16; First posted 2008-12-17 (Estimated); Last update posted 2011-08-30 (Estimated); Status verified 2011-08

CONDITIONS: Pregnancy
Keywords: preterm delivery; short cervical length; progesterone
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Active Comparator): previous preterm delivery, treatment with weekly injections of 17 alfa hydroxyprogesterone caproate.
  Interventions: Drug: 17 alfa hydroxyprogesterone caproate
- 2 (Active Comparator): previous preterm delivery, treatment with daily vaginal natural progesterone
  Interventions: Drug: natural progesterone
- 3 (Active Comparator): short cervical length, treatment with weekly injections of 17 alfa hydroxyprogesterone caproate.
  Interventions: Drug: 17 alfa hydroxyprogesterone caproate
- 4 (Active Comparator): short cervical length, treatment with daily vaginal progesterone 200 mg until 34 weeks gestation.
  Interventions: Drug: vaginal progesterone

INTERVENTIONS:
Drug: 17 alfa hydroxyprogesterone caproate — weekly injection of 250 mg until 34 weeks gestation
  Arms: 1
Drug: natural progesterone — previous preterm delivery, treatment with daily vaginal progesterone 200 mg until 34 weeks gestation.
  Arms: 2
Drug: 17 alfa hydroxyprogesterone caproate — weekly injection, 250 mg until 34 weeks gestation
  Arms: 3
Drug: vaginal progesterone — daily vaginal progesterone 200 mg until 34 weeks gestation.
  Arms: 4

SUMMARY:
Preterm deliveries play a significant role in neonatal morbidity and mortality. Previous studies showed that administration of progesterone to pregnant women at high risk, decrease spontaneous preterm deliveries.

The purpose of this study is to compare between two different modes of treatment with progesterone for the prevention of preterm delivery: weekly injection of 17 alfa hydroxyprogesterone caproate versus daily vaginal administration of progesterone in terms of efficacy, comfort and compliance, safety and cost of treatments.

ELIGIBILITY:
Inclusion Criteria:

* The subject has a history of spontaneous preterm delivery defined as earlier than 37 gestational week.
* The subject has a short cervical length defined as 25 mm before 24 weeks gestation.
* A singleton gestation.

Exclusion Criteria:

* Multifetal pregnancy.
* The subject has or will have a cervical cerclage in place.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2010-12; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
efficacy | 3 years

SECONDARY OUTCOMES:
comfort of use and consequently of that compliance | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Tal Biron-Shental, MD, Principal Investigator — Meir Medical Center, Israel, Affiliated to Tel Aviv University
Locations (1):
- Meir Medical Center, Kfar Saba, Israel